CLINICAL TRIAL: NCT07194967
Title: Effectiveness of Virtual Reality (HypnoVR) in Pain and Anxiety Management During Labor: Multicenter Randomized Controlled Trial
Brief Title: Virtual Reality for Pain and Anxiety Relief in Labor
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Collaborators: HypnoVR (Industry)
Responsible Party: Principal Investigator, Nesrine Souayeh, Associate Professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 02/2025
Record Dates: First submitted 2025-08-03; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Labor Pain; Anxiety
Keywords: Virtual Reality; hypnosis; pain management; anxiety; labor; Randomized Controlled Trial
MeSH Terms: conditions — Labor Pain; Anxiety Disorders; Agnosia

STUDY DESIGN:
Intervention Model Description: Parallel Randomized Controlled Trials
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The patients included in this arm received standard care with no additional intervention
- VR-group (Experimental): Patients in the intervention arm received standard obstetric care in addition to a virtual reality hypnosis session using the HypnoVR headset. The VR session, administered during the latent or active phase of labor, included immersive audiovisual content designed to promote relaxation, reduce anxiety, and alleviate pain through guided breathing and hypnotic suggestions
  Interventions: Device: Virtual Reality Hypnosis for Labor Pain and Anxiety Management

INTERVENTIONS:
Device: Virtual Reality Hypnosis for Labor Pain and Anxiety Management — For patients randomized to the intervention arm, the investigator will provide a clear explanation of the procedure and the use of the HypnoVR virtual reality headset. The investigator will remain present throughout the session to supervise the experience, using the companion tablet to monitor the visualization in real time.
  Participants will be invited to select one of eight immersive visual environments designed to promote relaxation and analgesia during labor. Available options include: Tropical Beach, Underwood, Underwater Dive, Zen Garden, Astral Travel, Winter Landscape, Aurora Borealis, and Oasis.
  Patients will be informed that they may discontinue the use of the headset at any time and for any reason, without any consequences for their standard medical care.
  Arms: VR-group

SUMMARY:
The aim of this study is to evaluate the impact of virtual reality hypnosis technique on pain and anxiety of women during labor. We will perform a randomized controlled trial on a group of labouring women at several hospitals in Tunis. We will also evaluate the satisfaction of women after the exposure to the virtual reality headset.

DETAILED DESCRIPTION:
This multicenter randomized controlled trial evaluates the effectiveness of a virtual reality hypnosis device (HypnoVR) in managing pain and anxiety during labor. Women in the latent and active phases of labor will be randomly assigned to either a VR intervention group or a control group receiving standard care.

Primary outcomes include pain level, measured using the Visual Analogue Scale (VAS), and anxiety level, assessed with the State-Trait Anxiety Inventory (STAI-Y). Both will be evaluated before and after the intervention.

Secondary outcomes include maternal vital signs (blood pressure and pulse), labor parameters (contraction frequency, duration, and intensity via NST), fetal parameters (heart rate and decelerations via Doppler), and maternal satisfaction (measured postpartum using a VAS satisfaction scale).

This study aims to determine whether HypnoVR can be an effective non-pharmacological method for improving the labor experience.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for inclusion in the study:

* Female participants aged between 18 and 45 years
* Primiparous or multiparous
* Singleton pregnancy
* Cephalic (vertex) presentation
* Gestational age between 37 and 41 completed weeks
* Admitted in spontaneous (uninduced) labor
* Low-risk pregnancy with no obstetric complications (e.g., no preeclampsia, gestational diabetes, or intrauterine growth restriction)
* Spontaneous and uneventful course of pregnancy
* At least four documented prenatal care visits during pregnancy
* Expressed desire for vaginal delivery
* Provided written informed consent to participate in the study

Exclusion Criteria: Participants will be excluded from the study if they meet any of the following criteria:

* History of any psychiatric disorder (e.g., anxiety, depression, bipolar disorder, psychosis, delirium) organic brain disease, or cognitive/developmental disorders)
* History of seizures or epilepsy
* Any degree of hearing impairment
* Any visual impairment
* History of face, neck, or head injuries that may interfere with the use of virtual reality equipment
* History of motion sickness or vestibular disorders (e.g., dizziness, vertigo)
* Chronic pain conditions or frequent migraines
* History of claustrophobia
* High-risk pregnancy (e.g., fetal growth restriction, placenta previa, or other significant maternal-fetal complications)
* Known fetal anomalies or placental abnormalities
* Labor pain not attributed to uterine contractions
* Induced labor (medically or pharmacologically initiated)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
pain level | Immediately before starting the intervention and immediately after completing the intervention
  The investigator assessed the pain level before and after the intervention using a Visual Analogue Scale VAS. The score ranges from 0 (no pain at all) to 10 (the worst pain imaginable).
anxiety level | Immediately before starting the intervention and immediately after completing the intervention
  The investigator assessed the Anxiety level using the State Trait Anxiety Inventory (STAI) forme Y. The score ranges from 20 to 80 and higher scores are associated with higher levels of anxiety.

SECONDARY OUTCOMES:
Blood pressure | Immediately before starting the intervention and immediately after completing the intervention, both systolic and diastolic blood pressures are mesures in millimetres of mercury (mmHg)
  Blood pressure in millimetres of mercury (mmHg)
Pulse rate | Immediately before starting the intervention and immediately after completing the intervention
  pulse rate mesured in heart beat per minute (bpm)
contractions intensity | Immediately before starting the intervention and immediately after completing the intervention
  contractions intensity is measured by NST machine, in millimiter of mercury (mmHg)
Contraction frequency | Immediately before starting the intervention and immediately after completing the intervention
  Contraction frequency per 10 mn These measurements were made using an NST machine
Contraction duration | Immediately before starting the intervention and immediately after completing the intervention
  contraction duration measured in minutes
Patient's satisfaction | After giving birth postpartum within two hours (H2)
  Satisfaction will be assessed using the Visual Analog Scale for Satisfaction (VAS; 0 = not at all satisfied, 10 = completely satisfied), with higher scores indicating greater satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Arous regional Hospital, Ben Arous, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) will not be shared due to concerns regarding participant confidentiality and data privacy. Although data will be collected in a de-identified format, the risk of re-identification cannot be completely eliminated, especially in small or vulnerable populations. In addition, no explicit consent for data sharing beyond the scope of the current study has been obtained from participants. Therefore, to comply with ethical standards and data protection regulations (e.g., GDPR), IPD will not most likely be made publicly available.

REFERENCES:
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Orhan M, Bulez A. The Effect of Virtual Reality Glasses Applied During the Episiotomy On Pain and Satisfaction: A Single Blind Randomized Controlled Study. J Pain Res. 2023 Jun 29;16:2227-2239. doi: 10.2147/JPR.S412883. eCollection 2023. PMID 37404226
- [Background] Slater M. Immersion and the illusion of presence in virtual reality. Br J Psychol. 2018 Aug;109(3):431-433. doi: 10.1111/bjop.12305. Epub 2018 May 21. PMID 29781508